CLINICAL TRIAL: NCT01102933
Title: RElevance of Biomarkers for Future Risk of Thromboembolic Events in UnSelected Post-myocardial Infarction Patients - an Observational Study (REBUS)
Brief Title: RElevance of Biomarkers for Future Risk of Thromboembolic Events in UnSelected Post-myocardial Infarction Patients
Acronym: REBUS
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: U-09-003
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for analysis of biomarkers and platelets. At the first visit after the hospital stay blood for DNA analysis will also be collected.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Unselected post-myocard infarct patients: Patients diagnosed with MI at Uppsala University Hospital

SUMMARY:
The study is an open, single center, observational study at the Cardiology Dept at Uppsala University Hospital. The number of patients included will be 410. The objectives are to:

Evaluate biomarkers and change of these related to myocardial infarction, during two years follow-up in an unselected patient population with a recent myocardial infarction.

Evaluate if an early change of biomarkers can be related to death, new myocardial infarction, and ischemic stroke in the same population after two and five years follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Myocardial infarction diagnosed by dynamic raised troponin I with at least one value above 0.1 µg/L. Together with at least one of the criteria; symptoms suggestive for myocardial infarction or development of significant Q wave.
2. Treated at the Department of cardiology, Uppsala University Hospital.
3. Ability to attend the scheduled visits for evaluation procedures.
4. Signed Informed Consent.

Exclusion Criteria:

1. Death ≤ 5 days after the myocardial infarction.
2. Not belonging to the catchment area of Uppsala University Hospital.
3. Lack of suitability for participation in the trial, for any reason, as judged by the Investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed wilth myocardial infarction and hospitalized at the Cardiology Department, Uppsala University Hospital, the study population will be unselected.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2010-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Death, myocardial infarction, stroke | Five years from study start
  Death: Death will be sub-classified by vascular or non-vascular primary cause. All deaths with unknown/uncertain cause will be categorized as vascular death.
  Myocardial Infarction(MI): Rehospitalization due to new non fatal MI or development of significant Q-wave.
  Stroke: Diagnosed as abrupt onset of focal neurological deficit persisting more than 24 hours.

SECONDARY OUTCOMES:
Venous thromboembolism, Arterial embolism, Bleeding | Five years from study start
  Venous thromboembolism: Deep venous thrombosis has to be diagnosed by ultrasonography or venography. Pulmonary embolism has to be diagnosed by spiral CT scan, pulmonary angiogram or ventilation-perfusion scanning.
  Arterial embolism: Diagnosed as an arterial event. Radiological evidence includes imaging studies.
  Bleedings: Classified as major or minor using International Society on Thrombosis and Haemostasis (ISTH). Major bleeds will be diagnosed as fatal and/or symptomatic bleeding in critical area or organ and/or bleeding associated with a decrease in Hb of 20 g/L or more or leading to transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Christersson, MD PhD, Principal Investigator — Cardiology Department, Uppsala University Hospital
Locations (1):
- Cardiology Department, Uppsal University Hospital, Uppsala County, Sweden